CLINICAL TRIAL: NCT01942486
Title: Thin Film Spectacle Coatings to Reduce Light Sensitivity and Headaches in Child and Adolescent Patients With Migraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Primary Children's Hospital (Other)
Responsible Party: Principal Investigator, Bradley Katz, M.D., University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00065178
Record Dates: First submitted 2013-06-14; First posted 2013-09-16 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Migraine Disorders; Photophobia
Keywords: migraine; photophobia; light sensitivity; melanopsin cells; intrinsically photosensitive retinal ganglion cells
MeSH Terms: conditions — Migraine Disorders; Photophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational Coating (Experimental)
  Interventions: Device: Investigational Coating

INTERVENTIONS:
Device: Investigational Coating

SUMMARY:
The purpose of this study is to determine if a special coating, applied to the surface of glasses can reduce the frequency and severity of migraine headaches in children and adolescents. This study is being conducted by researchers at Primary Children's Medical Center, The John Moran Eye Center, and the University of Utah Department of Electrical Engineering. The investigators have determined that a specific frequency of light is particularly bothersome to migraine patients. The coating they've developed is designed to block this frequency of light. Very few treatments are approved for the treatment of childhood migraine. The investigators hope that these glasses will provide a safe way to improve headaches in children.

ELIGIBILITY:
Inclusion Criteria:

1. Must be diagnosed with migraine with aura or migraine without aura
2. Must have at least 10 headache days per month

Exclusion Criteria:

1. Currently wearing a spectacle tint specifically prescribed for migraine or light sensitivity
2. Pregnant
3. Unwilling or unable in the judgment of the investigator to complete the study
4. Unavailable for any of the study visits
5. Light sensitive conditions: meningitis, iritis, blepharospasm, albinism
6. Degenerative diseases of the retina or optic nerve: diabetic retinopathy, ischemic optic neuropathy
7. Medications known to affect retinal or optic nerve function: hydroxychloroquine, chloroquine, ethambutol, amiodarone, erectile dysfunction drugs
8. Best corrected visual acuity less than 20/40 in either eye

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Katz, MD, Principal Investigator — University of Utah
Locations (1):
- Moran Eye Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational Coating: Subjects will wear an investigational coating on their glasses
Period: Overall Study
Arm/Group | Investigational Coating
Started | 35
Completed | 8
Not Completed | 27
Not completed — Lost to Follow-up | 27

BASELINE CHARACTERISTICS:
Groups:
- Investigational Coating: Investigational Coating
Arm/Group | Investigational Coating
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 35
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: HIT-6 Score
Description: The HIT-6 (Headache Impact Test) is a validated measure of the impact of headache on activities of daily living, functional health and well-being. The minimum score is 36 and the maximum score is 78. The higher the score, the more your headaches are adversely affecting activities of daily living. Patients who score higher than 50 are encouraged to seek help from their physician.
Time Frame: 12 weeks
Population: Only subjects that completed the trial were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Investigational Coating: Subjects will wear an investigational coating on their eyeglasses to reduce headache frequency
Arm/Group | Investigational Coating
Number analyzed (Participants) | 8
units on a scale | 62.3 (4.8)

ADVERSE EVENTS:
Time Frame: 3 years
Description: This was a minimal risk study with no risk of mortality and no risk of a serious adverse even
Groups:
- Investigational Coating: Subjects were asked to wear an investigational coating on their eyeglasses to reduce their headache severity
Arm/Group | Investigational Coating
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2013-07-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT01942486/Prot_002.pdf
  • Informed Consent Form: Parental Permission Form (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT01942486/ICF_000.pdf
  • Informed Consent Form: Assent Form (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT01942486/ICF_001.pdf